CLINICAL TRIAL: NCT02162212
Title: Diabetic Upper Extremity Pathophysiology, Limited Joint Mobility and Disability
Brief Title: Diabetic Shoulder Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014_DM_LJM; US NIH Grant R21 DK100793-01A1 (Other Grant/Funding Number: US NIH Grant)
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADA guideline Instructed (Active Comparator): The control intervention will be instruction in basic wellness activities according to the American Diabetes Association guidelines
  Interventions: Other: ADA Guideline Instructed
- Optimized Shoulder Movement Program (Experimental): The experimental intervention is the Optimized Shoulder Movement Program. Participants will be trained in a progressive home exercise program that includes passive stretching of end range shoulder flexion and external rotation, and active shoulder motion based on the participant's baseline "activity count" .
  Interventions: Other: Optimized Shoulder Movement Program

INTERVENTIONS:
Other: Optimized Shoulder Movement Program — A trained physical therapist will see the participant for a max of 6 visits over the 3 month intervention; for baseline instruction, and at 2, 4, 6, and 8 weeks to progress and check subject adherence before a final check-out and testing visit at 3 months. Participants will perform 3 assigned stretching motions a min of 2 sets of 10 reps each and will be instructed in active shoulder movements with a dose based on the subject's measured "activity count" at baseline and with enough duration to increase it by 10%. Exercise: 10-15 minutes 2x/day for 3 month duration. Participants will log their activity.
  Arms: Optimized Shoulder Movement Program
Other: ADA Guideline Instructed — The ADA guideline instructions are to include: blood sugar control (goal is A1c < 7.0%), physical activity (150 minutes/week of moderate intensity aerobic activity), foot care (examine feet daily, monofilament testing), and blood pressure control (goal is <130/80). Participants will receive a logbook to record daily outcomes. The goal of this intervention is to control for personal interactions with investigators and provide useful information for disease management but not provide intervention that likely would improve shoulder joint motion. The control group will be given instruction in the exercise program at the end of the 1 year study period.
  Arms: ADA guideline Instructed

SUMMARY:
The primary goal of this project is to determine how advanced glycation end-product (AGEs) accumulation and shoulder movement (humeral thoracic range of motion and "activity count") interact to contribute to shoulder limited joint mobility (LJM), pain and disability, and if an intervention consisting of a tailored dose of stretching and active shoulder movement can reduce these problems in people with diabetes mellitus (DM). The investigators will focus on the following measures that span health domains; Skin intrinsic fluorescence to measure AGEs; Ultrasound to measure supraspinatus tendon thickness; 3 dimensional joint range of motion and "activity counts" to measure shoulder movements; and the Disability of the Arm, Shoulder and Hand (DASH) questionnaire to measure patient reported pain and disability. The investigators will test the innovative hypothesis that metabolic and movement factors interact to cause severe shoulder problems in people with DM and that an optimized shoulder movement intervention can have an important impact on reducing the development of limited joint mobility, pain and disability in this population.

ELIGIBILITY:
Inclusion Criteria:

* individuals with type 2 DM and duration of diagnosed diabetes more than 10 years OR type 2 DM and presence of a 'positive prayer sign' OR shoulder flexion < 150 degrees; disability of arm, shoulder and hand (DASH) scores in the range of <70%; between the age of 40-70 will be recruited.

Exclusion Criteria:

* currently diagnosed adhesive capsulitis
* diagnosed rotator cuff tear
* recent (6 months) upper extremity injury and/or fractures
* surgery in the upper extremity or thorax
* cervical radiculopathy
* thoracic outlet syndrome
* stroke with residual upper extremity involvement
* severe skin allergies in area to be tested
* rheumatic conditions
* known connective tissue diseases
* carpal tunnel syndrome
* use of a cane
* individuals who engage in heavy upper extremity/ overhead use (ie, painters, tennis players) because they likely have a different mechanism of injury than those with low shoulder activity.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Arm elevation. | One year
  Arm elevation is a composite of shoulder (glenohumeral) and scapular motion and will be measured using goniometry and computer assisted kinematics. Glenohumeral elevation and external rotation motions are the main focus.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder, and Hand (DASH) questionnaire | One year
  The DASH is an established, standardized measure used to characterize pain and disability in the upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mueller, PT, PHD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Mueller MJ, Sorensen CJ, McGill JB, Clark BR, Lang CE, Chen L, Bohnert KL, Hastings MK. Effect of a Shoulder Movement Intervention on Joint Mobility, Pain, and Disability in People With Diabetes: A Randomized Controlled Trial. Phys Ther. 2018 Sep 1;98(9):745-753. doi: 10.1093/ptj/pzy070. PMID 29893977